CLINICAL TRIAL: NCT05456750
Title: The Investigation of Therapeutic Effect and Platelet Activity After Intravenous Laser Irradiation of Blood for Ischemic Stroke Patient
Brief Title: The Investigation of Therapeutic Effect and Platelet Activity After ILIB for Ischemic Stroke Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Liang-Cheng Chen, Principal Investigator, Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TSGH-D-111106
Record Dates: First submitted 2022-07-09; First posted 2022-07-13 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2024-07

CONDITIONS: Ischemic Stroke
Keywords: Ischemic Stroke; intravenous laser irradiation of blood; platele activity
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- treatment group (Experimental): The treatment group receive an intravenous helium-neon laser phototherapy. A vein indwelling needle will be placed in their veins located in the upper elbow, and the laser fiber catheter will be introduced through the indwelling cannula. The laser power is set between 2.5 ~ 3.0Mw, 60 minutes each time, once a day for five consecutive days each week, for 2 weeks (total 10 times in one course)
  Interventions: Device: Intravascular laser irradiation of blood
- control group (Sham Comparator): The steps for the control group are the same as the treatment group, except that the output power is adjusted to zero intensity.
  Interventions: Device: Intravascular laser irradiation of blood

INTERVENTIONS:
Device: Intravascular laser irradiation of blood — Low intensity intravenous laser irradiation of blood phototherapy is a method of a 632.8 nm red light penetrate into a vein through fiber and the brightness is 100 fold of the sun. The light accelerates blood and cells circulation in the human body, so that protein molecular structure would promote changes.

SUMMARY:
The aim of our study is to therapeutic effect and platelet activity after intravenous laser irradiation of blood for ischemic stroke patient

DETAILED DESCRIPTION:
Background : This research is designed through randomization, control, and double-blind trial to explore the clinical effectiveness of intravenous laser irradiation of blood for ischemic stroke patient; The research will further explore the changes in platelet activity after treatment. The light accelerates blood and cells circulation in the human body, so that protein molecular structure would promote changes. Pain control is indicated in such treatment, but still lacking evidence of neurological symptoms and functional improvement.

Purpose:This research is designed through randomization, control, and double-blind trial to therapeutic effect and platelet activity after intravenous laser irradiation of blood for ischemic stroke patient. Furthermore, to establish a new way of clinical rehabilitation therapy.

Method: The investigators plan to recruit 20 patients who are between the ages of 20 to 80 years old. The participants are required to have clear conscious and be able to communicate. The patient with mild to moderate stroke ( NIHSS=1-15), which onset between one month to 2 years will be included. The treatment group will receive an intravenous helium-neon laser phototherapy. A vein indwelling needle will be placed in their veins located in the upper elbow, and the laser fiber catheter will be introduced through the indwelling cannula. The power is set between 2.5 ~ 3.0Mw, 60 minutes each time, once a day for five consecutive days each week, for 2 weeks (total 10 times in one course). The steps for the control group are the same, except that the output power is adjusted to zero intensity. This plan will be explained to the patient in detail during the outpatient visit and patients will sign the consent form upon agreement. Before intravenous laser irradiation, three days, one month, and three months after the therapy, 20 ml of autologous peripheral venous blood need to be drawn for basic blood tests and platelet activity tests. At the same time, the clinical functions of patients will be evaluated, including NIHSS, mRS and Stroke Impact Scale (SIS).

ELIGIBILITY:
Inclusion Criteria:

* Aged between 20 to 80 years old
* Able to speak and understand Mandarin/Taiwanese
* No cognitive impairment
* Residual motor function impairment (mRS>1)
* Mild stroke (NIHSS=1-4) or Moderate stroke(NIHSS=5-15)
* No psychological disease

Exclusion Criteria:

* Severe stroke (NIHSS=16-42)
* History of intracerebral hemorrhage and other major surgery
* History of malignancy, chronic kidney disease
* Active infection
* Chronic hepatitis B or Chronic hepatitis C
* Unstable angina or acute myocardial infarction within 6 months
* Severe cognition impairment
* Pregnancy

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-07-28 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
National Institutes of Health Stroke Scale (NIHSS) | 3 month
  NIHSS is a measure of the severity of symptoms associated with ischemic stroke and is used as a quantitative measure of neurological deficit post stroke. NIHSS score is composed of 11 items, including consciousness, eye movement, visual fields, muscle power of four limbs, limbs ataxia, sensation, language, dysarthria and extinction. Each of which scores a specific ability between a 0 and 4. For each item, a score of 0 typically indicates normal function in that specific ability, while a higher score is indicative of some level of impairment. Total score are between 0-42.
  Measure before intravenous laser irradiation, three days, one month, and three months after the therapy.
Modified Rankin Scale (mRS) | 3 month
  The Modified Rankin Scale (mRS) is used to measure the degree of disability or dependence in the daily activities in patients who have had a stroke 0: No symptoms at all
  1. No significant disability despite symptoms; able to carry out all usual duties and activities
  2. Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance
  3. Moderate disability; requiring some help, but able to walk without assistance
  4. Moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance
  5. Severe disability; bedridden, incontinent and requiring constant nursing care and attention
  6. Dead Measure before intravenous laser irradiation, three days, one month, and three months after the therapy.
Stroke Impact Scale(SIS) | 3 month
  The Stroke Impact Scale (SIS) is a newly developed comprehensive outcome measure consists of items measuring 8 domains- strength, hand function, activities of daily living (ADL) and instrumental ADL, mobility, communication, emotion, memory and thinking, and participation. It was based on feedback from patients and their caregivers. Measure before intravenous laser irradiation, three days, one month, and three months after the therapy.

SECONDARY OUTCOMES:
Platelet activity | 3 month
  Platelet aggregation test. Measure before intravenous laser irradiation, three days, one month, and three months after the therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Liang-Cheng Chen, MD,MS, Principal Investigator — Department of Physical Medicine and Rehabilitation, Tri-Service General Hospital
Locations (1):
- Tri-service general hospital, Taipei, Taiwan